CLINICAL TRIAL: NCT00066625
Title: A Phase I and Pharmacokinetic Study of Oxaliplatin (Eloxatin™) in Combination With Bortezomib (PS-341, Velcade™) in Patients With Advanced Malignancy
Brief Title: Oxaliplatin and Bortezomib in Treating Patients With Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02552; NYU 02-12; N01CM62204 (NIH); CDR0000316444 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Oxaliplatin; Bortezomib

ARMS (1):
- Treatment (oxaliplatin, bortezomib) (Experimental): Patients receive oxaliplatin IV over 2 hours on days 1 and 15 and bortezomib IV over 3-5 seconds on days 1, 4, 15, and 18. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of oxaliplatin and bortezomib until the MTDs are determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  Interventions: Drug: oxaliplatin; Drug: bortezomib; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Phase I trial to study the effect on the body of combining oxaliplatin with bortezomib in treating patients who have metastatic or unresectable cancer. Drugs used in chemotherapy such as oxaliplatin use different ways to stop cancer cells from dividing so they stop growing or die. Bortezomib may stop the growth of cancer cells by blocking the enzymes necessary for tumor cell growth. Combining oxaliplatin with bortezomib may kill more cancer cells

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose and recommended phase II dose of oxaliplatin and bortezomib in patients with advanced malignancy.

II. Determine the dose-limiting toxicity of this regimen in these patients. III. Determine the toxicity profile of this regimen in these patients. IV. Determine the antitumor activity of this regimen in these patients. V. Determine the pattern of neurotoxicity and its reversibility in patients responding to prolonged administration of this treatment regimen.

VI. Determine whether the pharmacokinetics and pharmacodynamics of oxaliplatin or bortezomib are altered by the administration of the other agent in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive oxaliplatin IV over 2 hours on days 1 and 15 and bortezomib IV over 3-5 seconds on days 1, 4, 15, and 18. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of oxaliplatin and bortezomib until the maximum tolerated doses (MTDs) are determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed for at least 3 months.

PROJECTED ACCRUAL: A total of 15-30 patients will be accrued for this study within 4-15 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy for which standard curative or palliative measures do not exist or are no longer effective

  * Metastatic or unresectable disease
* No known brain metastases
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100
* More than 6 months
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin normal
* AST and ALT no greater than 5 times upper limit of normal
* Creatinine no greater than 1.5 mg/dL
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to any platinum or other study agents
* No pre-existing peripheral neuropathy
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other concurrent uncontrolled illness
* Prior thalidomide allowed provided patient has no clinical neuropathy
* Prior platinum or antitubulin agents allowed provided patient has no clinical neuropathy
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas and mitomycin) and recovered
* More than 3 weeks since prior radiotherapy and recovered
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational or commercial agents or therapies for the malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-07; Primary Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Probability of dose escalation according to true dose limiting toxicity (DLT) rate, based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v3.0 | Up to 28 days

SECONDARY OUTCOMES:
Area under the curve (AUC) estimates | Days 1 and 15 (course 1)
  Nonlinear compartmental analysis of the oxaliplatin pharmacokinetic data will be performed.
Pharmacodynamic assessments (20S proteasome inhibition data) | Days 1 and 15 (course 1)
  Summarized by dose and time using standard descriptive statistics. Asssessments will correlate the AUC in an Emax inhibitory model.
Sequence of drug administration in terms of PK interaction | Days 1 and 15 (course 1)
  AUC for oxaliplatin and 20-S proteasome inhibition will be calculated and compared for intra-patient variation using paired T-test.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Hochster, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States